CLINICAL TRIAL: NCT03387644
Title: Pregabalin Premedication for Conscious Sedation for Flexible Bronchoscopy: A Randomized Double Blind Controlled Study
Brief Title: Pregabalin Premedication for Conscious Sedation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Dr Ezzeldin Ibrahim, Assistant Professor in anaesthesia, intensive care, and pain medicine., Menoufia University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: MenoufiaU2015/5
Record Dates: First submitted 2017-12-15; First posted 2018-01-02 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Conscious Sedation
MeSH Terms: interventions — Pregabalin; Premedication

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregabalin (PG) (Active Comparator): Patients received 150 mg pregabalin one hour before the procedure.
  Interventions: Drug: Pregabalin (PG)
- Control placebo (C) (Placebo Comparator): Patients received placebo tablet one hour before surgery.
  Interventions: Drug: Control placebo (C)

INTERVENTIONS:
Drug: Pregabalin (PG) — Pregabalin 150 mg one hour before the procedure as premedication.
  Other Names: Pregabalin for premedication
  Arms: Pregabalin (PG)
Drug: Control placebo (C) — Placebo tablets one hour before the procedure as premedication.
  Other Names: Placebo for premeditation
  Arms: Control placebo (C)

SUMMARY:
Conscious sedation is usually required during flexible bronchoscopy. Sedation should be done without causing respiratory depression or loss of consciousness. The present study was designed to evaluate the advantage of pregabalin pre-medication on reducing sedatives and respiratory depression for patients undergoing flexible bronchoscopy with dexmedetomidine and midazolam.

DETAILED DESCRIPTION:
Seventy patients undergoing elective flexible bronchoscopy were randomly divided into two equal groups, 35 patients each. All patients received premedication one hour before the procedure. PG group received 150 mg pregabalin and C group received placebo. All patients sedated to achieve optimum working conditions. Intra-operative respiratory rate and post procedure patients' and pulmonologists' satisfaction were compared in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 21 and 65 years old American Society of Anaesthesiologists physical status II or III scheduled for elective flexible bronchoscopy

Exclusion Criteria:

* Patients with known allergy to any drug used in the study, chronic use of analgesics and/or sedatives, substance abuse, sleep apnea, renal or hepatic dysfunction, and psychiatric disorders.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-04-15 (Actual); Primary Completion 2016-11-24 (Actual); Study Completion 2017-05-16 (Actual)

PRIMARY OUTCOMES:
Total amount of sedative | 45 minutes during the procedure
  The total amount of the sedative used during the procedure.

SECONDARY OUTCOMES:
Patients' satisfaction | 30 minutes after the end of the procedure.
  Patient's satisfaction score was recorded using a score ranging from 0 not satisfied and 5 totally satisfied. The score was done using a questioner designed by the researchers.